CLINICAL TRIAL: NCT03035019
Title: Reducing Stress in Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Eva Szigethy, MD, Phd, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16040173
Record Dates: First submitted 2017-01-20; First posted 2017-01-27 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Stress
Keywords: anxiety; behavioral app
MeSH Terms: conditions — Anxiety Disorders | interventions — nano-lantern protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lantern for primary care patients (Experimental): All patients between the ages of 20-65 at specific primary care practices and score 5 or greater on the GAD7 questionnaire are offered the Lantern app to help with stress/anxiety.
  Interventions: Behavioral: Lantern

INTERVENTIONS:
Behavioral: Lantern — This pilot will evaluate how the availability of a virtual stress management resource can help patients reduce anxiety and improve quality of life.

SUMMARY:
Stress and anxiety can worsen quality of life in patients seen in primary care practices. This project is set in UPMC primary care practices (CMI) to evaluate how the availability of a virtual stress management program can help patients reduce stress and anxiety and improve their quality of life. The project will analyze the efficacy of the virtual stress management program at these practices so that it can then be utilized effectively in other medical settings where it can be offered as a part of clinical care to reduce stress and anxiety and improve the quality of life of medical patients who could benefit from a reduction in stress. This research is being piloted at these sites in the hopes of publishing results that show that it can be implemented in other practices throughout the country.

Additionally, at other UPMC CMI primary care sites, de-identified data will be collected in order to serve as a comparison.

DETAILED DESCRIPTION:
All patients who are receiving or seeking medical care at UPMC CMI practices are given the GAD7(anxiety) and SF-12(quality of life) as a part of their routine medical care. Since this project is occurring at the same practices where a randomized study evaluating treatments for acute back pain (IRB Protocol #015120249), patients with acute back pain will be excluded from this project.

Patient scores become part of the EMR (Epic). A best practice alert will be generated for patients in the age range of 20-65 (inclusive) and in the targeted GAD7 score range (GAD7 ≥5) to prompt the provider to recommend the stress management program (Lantern). The age range was chosen to exclude adolescents who may have different needs, and the geriatric population who is involved in other behavioral studies at these practices.

The Best Practice alert will prompt the clinic staff to gather promotional Lantern materials and pend an order in Epic for stress management registration. When the clinical staff sees the pended order and Lantern materials, clinic staff will decide if the stress management program is appropriate for the patient. The discussion will include a disclaimer that the stress management program does not offer treatment. Clinical staff and patient will also discuss whether or not the patient wishes to consent to participate in Lantern and be contacted Lantern. The clinical staff will question the patient about smartphone or tablet (specifically, iOS or Android) access/availability during the consent process. If the patient is interested, the clinician will submit the order and the patient will sign the consent to participate in the stress management program (Lantern). The use of Lantern is set up at these two CMI sites as part of this research study. It is not for normal clinical care for UPMC patients.

The order generates a paragraph about the stress management program provided to the patient as a written order. The order sends an Epic InBasket to the UPMC Enterprises project team (including the patient's MRN, name, date of birth and contact information). When each order is received, the UPMC Enterprises project team will enter the patient into the registration system, generating a unique ID for each patient.

The registration system will send out an email message to the third-party stress management program (including the unique ID, name, date of birth, and contact information) through a secure VPN connection between UPMC Enterprises and Lantern to inform them of people who have consented.

The third-party stress management program vendor, Lantern, will send a welcome message by email and text message to each patient consented by the UPMC research team. Patients also have the opportunity to directly sign up for Lantern while still in the primary care office.

Once the patient receives the welcome message by email or text, the patient can begin the program on a mobile device. Patients will be self-directed to complete modules of the stress management program.

Within 2-4 weeks after consent, a UPMC research team member will administer via phone a brief, approximately 10 minute questionnaire. This DSM5 cross-cutting measure level 1 is a validated screening tool capturing primary psychiatric conditions. The DSM5 will only be used for participants that score greater than or equal to 10 on the initial GAD7 in clinic or through MyUPMC. The techniques to try are available for users to access at any time. The coaches are not therapists, but are there to provide information and encouragement to the patient. To keep confidentiality, the coach only knows the first name of the patient. The coordinator of the coaches has access to the patient's identifying information if the patient has an escalation in distress/anxiety that needs to be addressed. This information will be passed to the PI when necessary as part of the escalation procedures (as outlined in the attachments - Escalation Procedure). The personally identifying information is held internally within the Amazon web services at Lantern. The coaches for the patients have access to an internal Coaching Portal where the coaches have a dashboard for each user. This dashboard includes all information that the user inputs into the Lantern program, including both direct messages to coaches and all content completed in the program. Coaches receive a notification when users complete a path in the program or send a message, which prompts a coach's response to the individual. Users will continue to self-monitor anxiety levels throughout the program after learning this skill in the first core component. (See Other Attachments - Example Messages from Lantern Coaches to read examples of how the coach interacts with the user as well as Sample Lantern Content.)

The 6 core components include:

1. Education and awareness about stress and how thoughts, emotions, and behaviors are interrelated. This provides the rationale of the cognitive-behavioral model. In this unit, patients will learn how to change thoughts and behaviors in order to change emotions.
2. Relaxation - patients learn several empirically supported relaxation techniques to manage stress/anxiety.
3. Thoughts - this unit is about the stories a person tells themselves and how these stories determine mood and help to decide what actions to take. This core component also guides patients on how to challenge assumptions about these thoughts/stories and how to create new stories.
4. Behavior Change and Exposure - patients will learn how to avoid things that contribute to stress and identify adaptive coping activities. Through learning the principle of exposure, patients learn how anxiety provoking situations can help to overcome anxiety in the long term.
5. Mindfulness - This unit is about taking a step back from thoughts and feelings to interrupt the thoughts-feelings-behaviors cycle. Several mindfulness exercises are offered so the patient can find the type that feels best.
6. Habit Formation/Maintaining Skills - Patients will reflect on what has been learned and work on making a habit out of the most effective techniques.

Lantern, the third-party program provider, will collect de-identified usage data (e.g., progression through the program, frequency of messages to coaches, and techniques completed) and quantitative data (e.g. self-monitoring anxiety score responses) as the patient progresses through the program. Lantern internally has a database that tracks user progress through the program, so Lantern can understand how patients have moved through the program. This de-identified data will be sent to the UPMC study staff coded only with the patient's unique ID.

Lantern will also generate usage data reports at regular intervals . The subject progression through Lantern is being fed into the research database from Lantern. These reports will also be coded by the patient's unique ID. The research team will send the usage progress report to EPIC to be included in the patient's medical record as a PDF.

At several time-points, Lantern will push self-reported validated questionnaires to patients enrolled in Lantern via a Qualtrics account. Lantern's Qualtric's account is a third party, HIPAA compliant survey tool. Thrive Network Inc. has a business associate agreement (BAA) with Lantern's Qualtric's account and owns all data collected through surveys.

Lantern's Qualtrics Account will push GAD7's and one additional item asking about satisfaction with the program to subjects. At 6 months post enrollment, participants at active (Lantern) sites will be sent a Qualtrics questionnaire with the GAD7, SF-12, Health Anxiety Sub-scale, Medical Utilization/Follow-up Questionnaire, and Patient Satisfaction questions. The purpose of the Health Anxiety Sub-scale is to evaluate how Health Anxiety changes may differ or are similar to GAD7 changes, and what impact both have on health care utilization.

In addition to the above assessment time points, patients will be pushed a GAD7 assessment via Qualtrics within one month of completing the Lantern program.

If the participant does not complete the Qualtrics survey at 6,and 12 months, the research team will contact the patient to prompt completion and offer to administer the measures over the phone. If a patient does not complete all of the modules of the Lantern program within a designated period of time, the patient will still be asked to fill out the questionnaires. In addition to these questionnaires, the research team will also access Epic records to understand medical utilization.

For this study, all patient responses through Lantern's Qualtrics account will be deidentified and stored within Lantern's Qualtrics account. Lantern will then share that deidentifed data with the UPMC clinical team using patient unique ID numbers. Lantern's coaches will not have access to any of the information collected via Qualtrics. Data from Qualtrics is pushed to the UPMC study database. GAD7 scores and participant program status will be sent in monthly enrollment reports to physicians and not be included as part of the electronic medical record (EPIC), unless a patient scores greater than or equal to 15, an In-Basket message is sent to the physician via Epic.

A secure database will be maintained within the UPMC firewall where all patient information will be de-identified. CARe will serve as the honest broker. Lantern will have access to Lantern's Qualtrics account - delivered surveys (tracked only by unique ID) but will not have access to any UPMC patient medical information.

A subset of patients (n=24) who were offered the Lantern program will be asked to participate in an in-depth qualitative telephone interview at 6 months after enrollment. Participants will be randomly selected and be balanced to include both those who completed or did not complete the program. The interviews will be completed by research staff contacting the randomly selected subjects. The qualitative interview will explore patient's experience with the program and areas of suggested improvement. All interviews will be audio-recorded and transcribed verbatim.

Comparison Sites: All patients who are receiving or seeking medical care at UPMC CMI comparison sites will not sign a consent form. Their information will be a medical record review of de-identified data in a limited dataset format from an honest broker.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are receiving or seeking medical care at UPMC CMI aged 20-65 who have a GAD7 score ≥ 5 must be English speaking and capable of understanding the informed consent and providing consent or assent and having access to a Smartphone.

Exclusion Criteria:

* Patients under age 20 and older than 65 will be excluded. Patients whose GAD7 score is <5 will also be excluded. Patients who do not own a smartphone or mobile device will also not be included. Since this project is occurring at the same practices where a randomized study evaluating treatments for acute back pain (IRB Protocol # 015120249), patients with acute back pain will be excluded from this project.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
GAD7 scores (anxiety) completion. | 12 months
  GAD7 anxiety questionnaires are completed at time points throughout the study
Patient satisfaction/acceptability post program | 6 months after consent
  A measure to determine patient satisfaction of the Lantern program

SECONDARY OUTCOMES:
Quality of life (SF-12) | 12 months
  SF-12 is a quality of life questionnaire participants complete.
medical utilization | 12 months
  Any medical treatment that occurred since consent, such as ER visits, # phone calls to practice, outpatient clinic visits and medical hospitalization days.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szigethy, MD, PHD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Szigethy E, Solano F, Wallace M, Perry DL, Morrell L, Scott K, Bell MJ, Oser M. A study protocol for a non-randomised comparison trial evaluating the feasibility and effectiveness of a mobile cognitive-behavioural programme with integrated coaching for anxious adults in primary care. BMJ Open. 2018 Jan 13;8(1):e019108. doi: 10.1136/bmjopen-2017-019108. PMID 29331971